CLINICAL TRIAL: NCT02263690
Title: Comparison of Three Different Anesthetic Approaches for Intravitreal Injections: A Prospective Randomized Trial
Brief Title: Comparison of Three Different Anesthetic Approaches for Intravitreal Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Retina Clinic, Sao Paulo, Brazil (Other)
Responsible Party: Principal Investigator, Gabriel Costa de Andrade, Gabriel Costa de Andrade, Retina Clinic, Sao Paulo, Brazil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RetinaC
Record Dates: First submitted 2014-09-30; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — proxymetacaine; Lidocaine; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group Drops (Active Comparator): proparacaine 0.5% drops (Group Drops)
  Patients from group Drops received a drop of proparacaine 0.5% before receiving a drop of povidone iodine 5%.
  Patients from Group Drops received a second drop of proparacaine 0.5%, 5 minutes after the drop of povidone iodine 5%.
  Interventions: Procedure: Group Drops
- Group SC (Active Comparator): proparacaine 0.5% drops plus subconjunctival lidocaine (Group SC)
  Patients from group SC received a drop of proparacaine 0.5% before receiving a drop of povidone iodine 5%.
  For the patients from Group SC, a subconjunctival bleb of anesthesia was created by injecting 0.4 ml of lidocaine 1% into the subconjunctival space, posteriorly to the superotemporal limbus with a 30-gauge, 1/2-inch needle attached to a 1-ml syringe.
  Interventions: Procedure: Group SC
- Group Gel (Active Comparator): Lidocaine gel 2% on the eye (Group Gel)
  Patients from Group Gel received 1 mL of 2% lidocaine gel on the eye before receiving the drop of povidone iodine 5%.
  For the patients from Group Gel, 1 mL of 2% lidocaine gel was applied on the eye before receiving the drop of povidone iodine 5%.
  Interventions: Procedure: Group gel

INTERVENTIONS:
Procedure: Group Drops — The patients in the group Drops received a drop of proparacaine 0.5% before receiving a peri-ocular drop of povidone iodide 5%. The patients in the group Drops received a second drop of proparacaine 0.5% 5 minutes after the drop of povidone iodide 5%
  Other Names: Proparacaine 0.5% drops
  Arms: Group Drops
Procedure: Group SC — The patients in the group SC received a drop of proparacaine 0.5% before receiving a peri-ocular drop of povidone iodide 5%. In the patients in the group SC, a subconjunctival bleb of anesthesia was created by injecting 0,4 mL of lidocaine 1% into the subconjunctival space 4 mm posterior to the superotemporal limbus with a 30-gauge, 1/2-inch needle attached to a 1-mL syringe.
  Other Names: Subconjunctival 1% Lidocaine
  Arms: Group SC
Procedure: Group gel — For the patients in group gel, the gel was placed on the eye before receiving the peri-ocular drop of povidone iodide 5%.
  Other Names: Lidocaine 2% gel
  Arms: Group Gel

SUMMARY:
92 patients in treatment with intravitreal injections were randomized to 1 of 3 groups: proparacaine 0.5% drops (Group Drops), proparacaine 0.5% drops plus subconjunctival lidocaine (Group SC), or 2% lidocaine gel (Group Gel). Patients were asked to score their pain experience using a visual analogue scale (VAS), a scale of 0 to 10, immediately following the injections as well as 10 minutes, 1 hour, 6 hours and 24 hours after. Patients also graded the overall injection experience as Excellent, Very Good, Fair, Poor or Awful. The physician evaluated the patient's eye movement during intravitreal injection in three levels: none or minimal (0), not compromising the injection (1), compromising the injection (2).

DETAILED DESCRIPTION:
This prospective, randomized, triple-armed trial compared the effectiveness of three different anesthetic approaches for intravitreal injections. Were included 92 consecutive patients scheduled to receive intravitreal injection of bevacizumab (Avastin, Genentech, Inc.) in one eye, from June 2014 to September 2014, evaluated at at a single center - Retina Clinic, Osasco, São Paulo, Brazil. The same ophthalmologist (CGA) administered both, anesthetic and therapeutic, injections. A masked nurse collected patient assessment responses and a masked statistician performed statistical analyses. The research followed the tenets of the Declaration of Helsinki and was approved by the Committee of Ethics in Research. All participants gave written informed consent prior to their participation.

Patients were randomized to 1 of 3 groups before injection: proparacaine 0.5% drops (Anestalcon®, Alcon Lab. do Brasil Ltda, São Paulo, Brazil), (Group Drops), proparacaine plus subconjunctival lidocaine 1% (Xylestesin®, Cristália, São Paulo, Brazil) (Group SC), or 2% lidocaine gel (Xylestesin®, Cristália, São Paulo, Brazil) (Group Gel).

A standardized method was used to prepare the injection site and disinfect the skin using povidone iodine 10%. Patients from groups Drops and SC received a drop of proparacaine 0.5% before receiving a drop of povidone iodine 5%. For the patients from Group Gel, the gel was placed on the eye before receiving the drop of povidone iodine 5%. Patients from Group Drops received a second drop of proparacaine 0.5%, 5 minutes after the drop of povidone iodine 5%. For the patients from Group SC, a subconjunctival bleb of anesthesia was created by injecting 0.4 ml of lidocaine 1% into the subconjunctival space, posteriorly to the superotemporal limbus with a 30-gauge, 1/2-inch needle attached to a 1-ml syringe. After 5 minutes of the drop of povidone iodine 5%, sterile field and a lid speculum were placed. The injection site was measured with calipers to be 3.5 mm or 4.0 mm posterior to the superotemporal limbus, for pseudophakic and phakic eyes, respectively. A 30-gauge 1/2-inch needle was used to inject 0.05 ml of bevacizumab (Avastin, Genentech, Inc.). After the injection, mild pressure was applied with a swabstick over the injection site to reduce vitreous reflux and subconjunctival hemorrhage another a drop of povidone iodine 5% was applied.

Immediately following the injection, a nurse, who was masked to the treatment, explained the 100-mm visual analog scale (VAS) for pain (Figure 1) and questioned the patients' level of pain perceived during the injection. This assessment was repeated 10 minutes, 1 hour, 6 hours and 24 hours later, without visualization of their prior responses. Patients were also asked to grade their overall experience with the injection procedure as Excellent (5), Very good (4), Fair (3), Poor (2) or Awful (1). The physician evaluated the patients' eye movement during intravitreal injection into three levels: none or minimal (0), not compromising the injection (1), compromising the injection (2). Complications that occurred during or after the procedures were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Indications for injection included neovascular AMD, DME and cystoid macular edema (CME) secondary to RVO.

Exclusion Criteria:

* Previous known allergic response to the topical anesthetics to be used.
* Previous intravitreal injections of drugs other than anti-VEGF agents
* Previous pars plana vitrectomy
* Anterior segment conditions that could affect pain sensation, such as conjunctival irritation, active conjunctivitis or keratitis or bullous keratopathy
* Patients using systemic analgesic or sedative medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pain experience and patient satisfaction after 3 different anesthetic approaches for intravitreal injections | immediately after injection, 10 minutes, 1 hour, 6 hours and 24 hours later
  Pain experience according the visual analogue scale (VAS), a scale of 0 to 10 (0 = no pain, 10 = worst pain ever).
  Patient satisfaction according the overall injection experience, graded by the patient as Excellent, Very Good, Fair, Poor, or Awful.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel C Andrade, M.D., Principal Investigator — Vitreo-retinal Fellow
Locations (1):
- Retina Clinic, Osasco, São Paulo, Brazil

REFERENCES:
- [Result] Aiello LP, Brucker AJ, Chang S, Cunningham ET Jr, D'Amico DJ, Flynn HW Jr, Grillone LR, Hutcherson S, Liebmann JM, O'Brien TP, Scott IU, Spaide RF, Ta C, Trese MT. Evolving guidelines for intravitreous injections. Retina. 2004 Oct;24(5 Suppl):S3-19. doi: 10.1097/00006982-200410001-00002. PMID 15483476
- [Result] Ulrich JN. Topical nepafenac after intravitreal injection: a prospective double-masked randomized controlled trial. Retina. 2014 Mar;34(3):509-11. doi: 10.1097/IAE.0b013e3182a0e611. PMID 23928675
- [Result] Brynskov T, Kemp H, Sorensen TL. No cases of endophthalmitis after 20,293 intravitreal injections in an operating room setting. Retina. 2014 May;34(5):951-7. doi: 10.1097/IAE.0000000000000071. PMID 24317292
- [Result] Nuzzi R, Tridico F. Local and systemic complications after intravitreal administration of anti-vascular endothelial growth factor agents in the treatment of different ocular diseases: a five-year retrospective study. Semin Ophthalmol. 2015 Mar;30(2):129-35. doi: 10.3109/08820538.2013.835833. Epub 2013 Oct 30. PMID 24171832
- [Result] Cintra LP, Lucena LR, Da Silva JA, Costa RA, Scott IU, Jorge R. Comparative study of analgesic effectiveness using three different anesthetic techniques for intravitreal injection of bevacizumab. Ophthalmic Surg Lasers Imaging. 2009 Jan-Feb;40(1):13-8. doi: 10.3928/15428877-20090101-05. PMID 19205490
- [Result] Kaderli B, Avci R. Comparison of topical and subconjunctival anesthesia in intravitreal injection administrations. Eur J Ophthalmol. 2006 Sep-Oct;16(5):718-21. doi: 10.1177/112067210601600509. PMID 17061223
- [Result] Bartfield JM, Holmes TJ, Raccio-Robak N. A comparison of proparacaine and tetracaine eye anesthetics. Acad Emerg Med. 1994 Jul-Aug;1(4):364-7. doi: 10.1111/j.1553-2712.1994.tb02646.x. PMID 7614283
- [Result] Blaha GR, Tilton EP, Barouch FC, Marx JL. Randomized trial of anesthetic methods for intravitreal injections. Retina. 2011 Mar;31(3):535-9. doi: 10.1097/IAE.0b013e3181eac724. PMID 21102369
- [Result] Davis MJ, Pollack JS, Shott S. Comparison of topical anesthetics for intravitreal injections : a randomized clinical trial. Retina. 2012 Apr;32(4):701-5. doi: 10.1097/IAE.0b013e31822f27ca. PMID 22282296
- [Result] Kozak I, Cheng L, Freeman WR. Lidocaine gel anesthesia for intravitreal drug administration. Retina. 2005 Dec;25(8):994-8. doi: 10.1097/00006982-200512000-00007. PMID 16340529
- [Result] Friedman SM, Margo CE. Topical gel vs subconjunctival lidocaine for intravitreous injection: a randomized clinical trial. Am J Ophthalmol. 2006 Nov;142(5):887-8. doi: 10.1016/j.ajo.2006.06.033. PMID 17056383
- [Result] Page MA, Fraunfelder FW. Safety, efficacy, and patient acceptability of lidocaine hydrochloride ophthalmic gel as a topical ocular anesthetic for use in ophthalmic procedures. Clin Ophthalmol. 2009;3:601-9. doi: 10.2147/opth.s4935. Epub 2009 Nov 2. PMID 19898665
- [Result] Boden JH, Myers ML, Lee T, Bushley DM, Torres MF. Effect of lidocaine gel on povidone-iodine antisepsis and microbial survival. J Cataract Refract Surg. 2008 Oct;34(10):1773-5. doi: 10.1016/j.jcrs.2008.05.056. PMID 18812132
- [Result] Inman ZD, Anderson NG. Incidence of endophthalmitis after intravitreal injection of antivascular endothelial growth factor medications using topical lidocaine gel anesthesia. Retina. 2011 Apr;31(4):669-72. doi: 10.1097/IAE.0b013e3181ef463d. PMID 21178659
- [Result] Charles S, Rosenfeld PJ, Gayer S. Medical consequences of stopping anticoagulant therapy before intraocular surgery or intravitreal injections. Retina. 2007 Sep;27(7):813-5. doi: 10.1097/IAE.0b013e318154b9f2. No abstract available. PMID 17891002
- [Result] Meyer CH, Callizo J, Mennel S, Kussin A. Perioperative management of anticoagulated patients undergoing repeated intravitreal injections. Arch Ophthalmol. 2007 Jul;125(7):994. doi: 10.1001/archopht.125.7.994. No abstract available. PMID 17620596